CLINICAL TRIAL: NCT05159570
Title: Modulation of Circulating Levels of the Ketone Body 3-hydroxybutyrate in Patients With Type 2 Diabetes and Heart Failure With Preserved Ejection Fraction: Metabolic Effects.
Brief Title: Modulation of Circulating Levels of the Ketone Body 3-hydroxybutyrate in Patients With Type 2 Diabetes and Heart Failure With Preserved Ejection Fraction: Metabolic Effects. (KETO-HFpEF-Metabolic)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00550
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Diabetes Mellitus, Type 2; Ketonemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone ester (Experimental)
  Interventions: Dietary Supplement: Ketone ester
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone ester — Commercially available ketone supplement
  Arms: Ketone ester
Dietary Supplement: Placebo drink — Isocaloric placebo
  Arms: Placebo

SUMMARY:
Heart failure (HF) is among the most common causes of death in patients with type 2 diabetes (T2D). Ketones, 3-hydroxybutyrate (3-OHB), have shown to have beneficial effects in patients with hearth failure with reduced ejection fraction. However, this have never been investigated in patients with heart failure with preserved ejection fraction (HFpEF).

In this study we would like to investigate the effect of 14 days modulation of circulating ketone body levels on whole body and skeletal metabolism in patients with HFpEF and T2D.

ELIGIBILITY:
Inclusion Criteria:

(i) Type 2 diabetes, (ii) LVEF > 40 %, (iii) a clinical diagnosis of HFpEF and/or left ventricular hypertrophy (posterior wall thickness > 12 mm) and/or previous myocardial infarction, (iiii) age ≥ 18 years old, and (iv) one of the following criteria (a-d) should be fulfilled:

Echocardiographic signs of diastolic dysfunction E/e' > 8 Septal e ́< 7 cm/s and/or lateral e ́ < 10 cm/s Left atrium volume index ≥34 mL/m2 and/or left atrial diameter > 4 cm NT-proBNP > 125 pg/ml.

Exclusion Criteria:

* Insulin treatment, inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Differences in lipolysis rate | After 14 days treatment
  Measured as differences in palmitate flux

SECONDARY OUTCOMES:
Changes in glucose kinetic | After 14 days treatment
  Measured by glucose tracer.
Changes in signaling in muscle and adipose tissue | After 14 days treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided